CLINICAL TRIAL: NCT01805102
Title: Preimplantation Factor (PIF): Biomarker Detection in Maternal Blood - Correlation With Live Birth.
Brief Title: Correlation Between PIF Maternal Serum Levels and Pregnancy Outcome
Acronym: PIFBlood1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BioIncept LLC (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: BioIncept LLC-2; GFI Merck Serono 2012 (Other Grant/Funding Number: GFI-1)
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Pregnancy
Keywords: In vitro fertilization; implantation; miscarriage; live birth
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — maternal blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- maternal serum: measurement by immunoassay

SUMMARY:
PIF: biomarker of pregnancy, miscarriage, premature birth, preeclampsia, placenta accreta.

Except for serum hCG, no pregnancy-complication markers are widely employed to predict the need for medical intervention. Since circulating PIF is present from very early and throughout viable pregnancy, it may represent a specific biomarker candidate. PIF levels will be analyzed in serum of pregnant women in a range of settings: a) following IVF; b) index pregnancy of women with history of recurrent pregnancy loss, c) index pregnancy of women with history of placenta mediated complications such as: intrauterine growth restriction, spontaneous idiopathic preterm delivery, and preeclampsia; and d) index pregnancy in women with evidence of abnormal placentation, namely placenta accreta and related conditions.

DETAILED DESCRIPTION:
We will assess PIF prospectively in maternal serum throughout viable pregnancy in order to assess its performance characteristics in predicting viability. More than 250 pregnancies after IVF will be studied as control patients. This PIF longitudinal pregnancy follow up will be compared to those observed for women at risk of pregnancy complications, those with previous such pregnancy.

One objective will be also to define PIF as a biomarker of pregnancy outcome. Then, we will also assess PIF levels in the maternal serum of women with pregnancy complications like miscarriage, preeclampsia, placenta accreta, preterm birth and intrauterine fetal growth restriction.

Our objective is to evaluate PIF maternal serum level in index pregnancy for women with previous pregnancy complications (miscarriage, preeclampsia, intrauterine fetal growth restriction, preterm birth) as listed above and consider at risk pregnancy complication recurrence. Data will be compared with control women (spontaneous pregnancy, singleton gestations, no medical treatment, normal delivery) and pregnant women with SET or MET after IVF.

Prospectively, we will include all patients with a previous pregnancy complications and 100 control women and 200 women after IVF cycles, over 36 months.

PIF assessment will be performed using specific antibody marked with a fluorescent dye, in Luminex® reader.

- PIF predictive value on pregnancy prognosis For all women, 5 routine blood draws will be conducted. The first one will occur after SET or MET (multiple embryo transfer) in women conceived via IVF and resulting in a successful ongoing pregnancy. Specifically, PIF levels in maternal serum will be evaluated 5 weeks after embryo transfer. In women with a history of previous pregnancy complication and control ones, a maternal blood draw will be obtained upon diagnosis of pregnancy, in the first trimester. The remainder of the blood draws (three per patient) will be obtained at the time of routine antenatal blood draws (typically 10-13 weeks for first trimester screening 15-20 weeks for MSAFP assessment; 24-28 wks for glucose screening and complete blood count).

If a complication will occur, a sixth blood draw will be done at the diagnosis time.

Definitions:

Preeclampsia is defined as hypertension (sustained elevations in systolic BP to at least 140 mmHg and/or in diastolic BP to at least 90 mmHg for at least 6 hours) in association with proteinuria (300 mg/24 hours) or concentration of at least 30 mg/dl (at least 1+ on dipstick) in at least 2 random urine samples collected at least 6 hours apart.

Intrauterine fetal growth restriction defined as a birth weight ≤10% percentile for gestational age, unrelated to malformations, karyotype abnormalities, obvious fetal infections or uterine malformations. IUGR will be ascertained from hospital records related to the current pregnancy.

Miscarriage, or fetal loss, is defined as the spontaneous loss of pregnancy prior to 20 weeks gestation, and recurrent pregnancy loss is defined as 2 or more failed pregnancies (documented by ultrasound or histological exam). Unexplained fetal death is defined as death ≥ 20 wks gestation unrelated to major malformations, karyotype abnormalities, maternal or fetal infections, maternal uterine or cervical malformations. Fetal death will be ascertained from hospital records related to the current pregnancy. The research nurse will complete a fetal death form, which will include information on autopsy results (if available), maternal serologies, toxicologies, maternal/fetal infections, uterine and cervical malformations, fetal/ placental karyotypes, isoimmunization.

Placenta accreta is defined as the direct apposition of placental villi to the myometrium. Placenta accreta is classified according to the degree to which the myometrium is penetrated by placental villi (KhongTY. J ClinPathol. 2008 Dec;61(12):1243-6).

Preterm birth is defined as a spontaneous birth occurring before 37 completed weeks of gestation, and at or after 20 weeks of gestation.

Methodology All women will be fully informed and a written consent to participate in the study will be duly obtained.

Maternal serum retrieval

Maternal serum will be collected during routine blood draw:

* at 5 weeks after embryo transfer for pregnant women after IVF, and for women with previous pregnancy complication upon the diagnosis of pregnancy in the first trimester (P1)
* at first trimester screening 10-13 wks (P2)
* at second trimester analyte screening, 15-20 wks (P3)
* at screening for diabetes, and anemia assessment 24-28 wks (P4)
* at admission for labor and delivery (P5)
* at pregnancy complication diagnosis (P6) PIF level evaluation As previously described Analysis Correlate PIF levels in maternal serum with pregnancy complications. Results of PIF detection on maternal serum will be correlated to pregnancy outcome, and pregnancy complications. Evolution of PIF level during pregnancy will be also evaluated. Controls will be matched for parity, multiple gestation and gestational age of blood draw (+/- 2wks).

Statistical analysis plan components, (no template provided) URC Paris Ile de France Ouest As pregnancy complications occurred in 25% of cases, patient number has been estimated to be 1350. 350 pregnancy complications will occur during the study.

The sample size will provide a 5% precision for a 30% event occurrence with a 5% standard deviation.

ELIGIBILITY:
Inclusion criteria:

* Women attending a perinatal center who are properly informed and willing to participate in this study. Women included in the participating center with previous pregnancy complication and pregnant women after IVF (SET or MET). PIF levels evaluation in maternal serum (P1 to 5) will be evaluated for all pregnant women.

Exclusion criteria:

* Women who will refuse to participate in the program.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women followed during pregnancy in perinatal centers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Maternal serum PIF levels correlation with pregnancy viability | up to 12 weeks
  Maternal blood will be collected serially following implantation. PIF levels will be recorded. Patients will be followed by standard methods including blood tests and ultrasound until viability is established. Implantation failure (ie chemical pregnancy) miscarriage, evidence of gestational sac will be recorded.

SECONDARY OUTCOMES:
Compare pregnancy outcome to low/high PIF levels in maternal blood | up to live birth
  PIF levels will be correlated with low and high risk pregnancy events. Once viability is established then patients will be monitored a) following IVF; b) index pregnancy of women with history of recurrent pregnancy loss, c) index pregnancy of women with history of placenta mediated complications such as: intrauterine growth restriction, spontaneous idiopathic preterm delivery, and preeclampsia; and d) index pregnancy in women with evidence of abnormal placentation, namely placenta accreta and related conditions until eventual delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Eytan R Barnea, MD, Study Chair — BioIncept LLC
Locations (5):
- Yale Women and Children's Center for Blood Disorders & Yale Fertility Center, New Haven, Connecticut, United States
- France (3):
  - Poissy St Germain Hospital, Poissy, Cedex
  - Lab Clement - Seine St Denis Hospital, Le Blanc Mesnil, Paris
  - Versailles St Quentin University, Poissy
- Helena Venizelou Hospital, Athens, Greece